CLINICAL TRIAL: NCT03985345
Title: Prospective Evaluation of the Connected EMY Biofeedback Probe in the Management of Stress Urinary Incontinence.
Acronym: Reduc@home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: FIZIMED (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6990
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EMY Probe (Experimental)
  Interventions: Device: intravaginal device (probe) EMY

INTERVENTIONS:
Device: intravaginal device (probe) EMY — Free use of EMY and its mobile application for 10 minutes during 5 different days per week.

SUMMARY:
After birth, the perineum has to be trained in order to recover its functions.

This study is designed to assess the quality of life evolution with the EMY connected device.

The secondary purposes are to evaluate patient compliance to the EMY probe, to observe the evolution of urine scores over the duration of the trial in order to consider a comparative study thereafter, and to evaluate the interest of using the EMY connected perineal probe in the context of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Women with urinary leakage, at least once a week or more since more than 3 months
* Women aged 18 and over, no upper age limit
* Patient having given birth since 6 months minimum
* Patient able to do an effective voluntary contraction and avoiding abdominal synergy and apnea during contraction (attested by the health professional partner who leads the patient to the study)
* Patient who has responded favorably to a perineal reeducation with at least 2 sessions (attested by the health professional partner who leads the patient to the clinical study), rehabilitation of stress urinary incontinence or mixed incontinence with predominance of stress urinary incontinence
* Signed informed consent form
* Effective contraception throughout the study (declarative)
* The patient must have a smartphone running at least the Android 5 and iOS 8 versions
* The patient must know how to read and write French

Exclusion Criteria:

* Patient practicing any other perineal reeducation during the study period
* Patient with neurological disease or congenital malformation, urinary incontinence or prolapse treated surgically or medically or perineal hypoesthesia or local conditions that prohibit the use of an intravaginal device
* Patient with an urge urinary incontinence or mixed urinary incontinence with a predominance of urgency.
* Contraindication to the use of the medical device
* Patient with Genito-urinary cancer (in the last 5 years)
* Patient with extra-uretral "incontinence" (fistula, ectopic ureter)
* Patient with severe urinary retention
* Patient carrying a sacral neuromodulation case
* Subject in exclusion period (determined by previous or current study)
* Impossibility to give the patient clear information (patient in emergency situation, patient with difficulties for understanding, ...)
* Patient under the protection of justice
* Patient under guardianship or curatorship
* Pregnancy (positive urine test)
* Breastfeeding patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

PRIMARY OUTCOMES:
Contilife questionnaire | The change of the quality of life will be assessed : completion of Contilife questionnaire at the inclusion visit (Day 0), one month after inclusion visit (Month1), 2 months after inclusion visit (Month2) and 3 months after inclusion (Month3).
  A quality of life questionnaire will be used to follow the quality of life evolution for patients with stress urinary incontinence (UI) using the EMY device.

SECONDARY OUTCOMES:
The patient compliance to the EMY device | Patients will complete the tracking notebook each time they use the EMY device during 3 months of the clinical research study (from inclusion, until visit Month3).
The urinary scores | The change in the urinary scores will be assessed. The ICIQ-SF questionnaire will be completed by patients at the inclusion visit (Day0) and on visits Month1, Month2 and Month3.
The interest of using the EMY connected perineal device in the context of stress urinary incontinence | The PGI-I questionnaire will be completed at visit Month3 (3 monhs after inclusion visit).
The interest of using the EMY connected perineal device in the context of stress urinary incontinence | The questionnaire of interest will be completed at visit Month3 (3 monhs after inclusion visit).

CONTACTS AND LOCATIONS:
Locations (1):
- Strasbourg University Hospitals, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jochum F, Garbin O, Godet J, Ragueneau M, Meyer C, Billecocq S, Lecointre L, Akladios C, Host A. Prospective evaluation of the connected biofeedback EMY Kegel trainer in the management of stress urinary incontinence. J Gynecol Obstet Hum Reprod. 2022 Feb;51(2):102280. doi: 10.1016/j.jogoh.2021.102280. Epub 2021 Dec 1. PMID 34861424